CLINICAL TRIAL: NCT02635061
Title: A Phase 1b Study of the Selective HDAC6 Inhibitor ACY-241 in Combination With Nivolumab in Patients With Unresectable Non-Small Cell Lung Cancer
Brief Title: Selective HDAC6 Inhibitor ACY 241 in Combination With Nivolumab in Patients With Unresectable Non Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-ST-203
Record Dates: First submitted 2015-12-14; First posted 2015-12-18 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — citarinostat; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ACY-241 in combination with nivolumab (Experimental)
  Interventions: Drug: ACY-241; Drug: Nivolumab

INTERVENTIONS:
Drug: ACY-241 — Specified dose on specified days
Drug: Nivolumab — Specified dose on specified days
  Other Names: Opdivo

SUMMARY:
Determine the safety, tolerability, dose limiting toxicities (DLTs), and maximum tolerated dose (MTD) of ACY 241 in combination with nivolumab.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand and voluntarily sign an informed consent form (ICF).
2. Must be ≥ 18 years of age at the time of signing the ICF.
3. Must be able to adhere to the study visit schedule and other protocol requirements.
4. Patients must have histologically confirmed unresectable NSCLC for which nivolumab is clinically appropriate. Patients must have had one line of prior therapy and have progressed or have discontinued due to toxicity.
5. Measurable disease by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) and Immune related Response Criteria (irRC).
6. Life expectancy > 12 weeks.
7. Must have Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
8. Willingness to have pre treatment and on treatment tumor biopsies.
9. Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Female patients of childbearing potential must agree to use adequate contraceptive measures until 3 months after the last study drug is taken. Females of childbearing potential must have a negative pregnancy test. It is not known if the antideacetylase activity of this experimental drug may be harmful to the developing fetus or nursing infant.
10. Male patients should be willing to use barrier contraceptive (ie, condoms) until 3 months after last study drug is taken.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from giving informed consent.
2. Any serious concurrent medical conditions, laboratory abnormality, or psychiatric illness that might make the patient nonevaluable, put the patient's safety at risk, or prevent the patient from following the study requirements.
3. Pregnant or lactating females.
4. Patients with uncontrolled brain metastases. Existing brain metastases must have been previously treated and currently stable.
5. Patients who have had chemotherapy within 14 days before entering the study or those who have not recovered from AEs to ≤ Grade 1 due to agents administered more than 14 days earlier.
6. Previous therapy with histone deacetylase (HDAC) inhibitor and/or anti PD 1, anti PD L1, or anti CTLA4 immunotherapy.
7. Any of the following laboratory abnormalities:

   * ANC < 1,500/µL
   * Platelet count < 100,000/µL
   * Hematologic growth factors are not allowed at Screening or during the first cycle of treatment
   * Hemoglobin < 9 g/dL (< 5.5 mmol/L; previous red blood cell transfusion is permitted)
   * Creatinine > 1.5 × upper limit of normal (ULN)
   * AST or ALT > 2.5 × ULN. For patients with liver metastasis AST or ALT > 5 × ULN
   * Serum total bilirubin > 1.5 mg/dL or > 3 × ULN for patients with hereditary benign hyperbilirubinemia
8. Corrected QT interval (QTc) using Fridericia's formula (QTcF) value > 480 msec at Screening; family or personal history of long QTc syndrome or ventricular arrhythmias including ventricular bigeminy at Screening; previous history of drug induced QTc prolongation or the need for treatment with medications known or suspected of producing prolonged QTc intervals on electrocardiogram (ECG).
9. Congestive heart failure (New York Heart Association Class III or IV), myocardial infarction within 12 months before starting study treatment, or unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris.
10. Patients with chronic autoimmune disease(s) requiring systemic immunosuppression.
11. Positive human immunodeficiency virus, hepatitis B virus, and hepatitis C virus infection.
12. Patients who received any of the following within the 14 days before initiating study treatment: major surgery, radiation therapy, and/or systemic therapy (standard or an investigational or biological anticancer agent).
13. Current enrollment in another clinical study involving treatment and/or is receiving an investigational agent for any reason, or use of any investigational agents within 14 days of initiating study treatment.
14. Incidence of gastrointestinal disease that may significantly alter the absorption of ACY 241.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | one to two years
recommended Phase 2 dose (RP2D) of ACY 241 in combination with nivolumab | one to two years

SECONDARY OUTCOMES:
preliminary antitumor activity of ACY 241 in combination with nivolumab | one to two years
Maximum Plasma Concentration [Cmax] of ACY 241 in combination with nivolumab on biomarkers in peripheral blood and tumor tissue | one to two years

CONTACTS AND LOCATIONS:
Overall Officials: Ileana Elias, MD, Study Director — Celgene
Locations (1):
- Local Institution - 350, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Awad MM, Le Bruchec Y, Lu B, Ye J, Miller J, Lizotte PH, Cavanaugh ME, Rode AJ, Dumitru CD, Spira A. Selective Histone Deacetylase Inhibitor ACY-241 (Citarinostat) Plus Nivolumab in Advanced Non-Small Cell Lung Cancer: Results From a Phase Ib Study. Front Oncol. 2021 Sep 6;11:696512. doi: 10.3389/fonc.2021.696512. eCollection 2021. PMID 34552864
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome